CLINICAL TRIAL: NCT00993343
Title: A Prospective Randomized Study Comparing Rapamune and Tacrolimus vs. Cyclosporine and Methotrexate as Immune Prophylaxis in Allogeneic Hematopoietic Stem Cell Transplantation, Using HLA-A, -B, -DRβ1 Identical Related or Unrelated Donors. A Nordic Multicenter Study.
Brief Title: Randomized Trial Comparing Sirolimus and Tacrolimus Versus Cyclosporine and Methotrexate as Graft-versus-host Disease (GVHD) Prophylaxis After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jonas Mattsson, Medical Director, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 070101
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Graft-versus-host Disease; Survival
Keywords: GVHD; tacrolimus; sirolimus; cyclosporine; allogeneic; stem cell transplantation; Relapse-free survival
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sirolimus; Tacrolimus; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine + Methotreaxte (Active Comparator)
  Interventions: Drug: cyclosporine/methotrexate
- sirolimus + tacrolimus (Active Comparator)
  Interventions: Drug: Sirolimus/tacrolimus

INTERVENTIONS:
Drug: Sirolimus/tacrolimus — Standard GVHD prophylaxis
  Arms: sirolimus + tacrolimus
Drug: cyclosporine/methotrexate — Standard GVHD prophylaxis
  Arms: Cyclosporine + Methotreaxte

SUMMARY:
To evaluate if rapamune + tacrolimus immunosuppressive prophylaxis is better than the established therapy using cyclosporine and methotrexate, a Nordic prospective multicenter randomized study will be performed. Patients will be randomized to treatment with rapamune combined with tacrolimus, or the established therapy using cyclosporine and methotrexate.

DETAILED DESCRIPTION:
Primary endpoint The primary endpoint is grade II-IV acute GVHD in the two groups. GVHD is diagnosed clinically and graded from 0 to IV. The diagnosis is clinical and biopsies from skin, liver and gut is used according to the routines at each participating center.

Other study parameters

1. Time to neutrophils >0.5 x 109/L.
2. Time to platelets >20 x 109/L and 50 x 109/L.
3. Platelet level 30 days after transplant.
4. Transfusion requirements of platelets, erythrocytes, granulocyte transfusions during the first 30 days.
5. Non-engraftment (graft failure/rejection).
6. Grade of acute GVHD.
7. Incidence of chronic graft-versus-host disease graded as limited or extensive and mild, moderate and severe.
8. Transplant-related mortality.
9. Probability of relapse in patients with haematological malignancies.
10. Survival.
11. Relapse-free survival.
12. Infections by bacteria, virus and fungi. Cytomegalovirus reactivation is also followed by PCR.
13. Side-effects. Side-effects regarding hematopoiesis, liver test, renal function, cardiac function, neurology, endocrinology, etc., are taken from the patients' charts. These parameters are followed regularly after transplantation.

Inclusion criteria Chronic myeloid leukemia (CML) in 1st or 2nd chronic phase, acute myeloid leukemia (AML) in complete remission, acute lymphoblastic leukemia (ALL) in complete remission, myelodysplastic syndrome, chronic lymphocytic leukemia, lymphoma, non-malignant disorders, severe aplastic anemia, hemoglobinopathies and metabolic disorders

ELIGIBILITY:
Inclusion Criteria:

* Chronic myeloid leukemia (CML) in 1st or 2nd chronic phase, acute myeloid leukemia (AML) in complete remission, acute lymphoblastic leukemia (ALL) in complete remission, myelodysplastic syndrome, chronic lymphocytic leukemia, lymphoma, non-malignant disorders, severe aplastic anemia, hemoglobinopathies and metabolic disorders

Exclusion Criteria:

* Recipients of major HLA-mismatched grafts.
* Patients who are addicted to drugs or alcohol.
* Patients who receive other stem cell source than bone marrow or peripheral stem cells, for instance cord blood transplants.
* Patients with relapse or blast crisis of their malignant disease.
* Prior allogeneic transplant using any hematopoietic stem cell source
* Seropositive for the human immunodeficiency virus (HIV)
* Uncontrolled bacterial, viral, or fungal infection (progression of clinical symptoms) Pregnant (positive serum human chorionic gonadotropin [β-HCG] test) or breastfeeding within 4 weeks of study entry
* Kidney function: serum creatinine outside the normal range for age, or measured creatinine clearance less than 40 mL/min/1.72m² within 4 weeks of study entry and proteinuria >0.3 g/day
* Liver function: most recent direct bilirubin, ALT, or AST greater than two times the upper limit of normal within 4 weeks of study entry
* Lung disease: in adults, FVC or FEV1 less than 60% of predicted value (corrected for hemoglobin); in children, overt hypoxemia, as measured by an oxygen saturation of less than 92% within 4 weeks of study entry
* Cardiac ejection fraction of less than 45% in adults and children, or less than 26% shortening fraction in children within 4 weeks of study entry
* Cholesterol level greater than 300 mg/dL or triglyceride level greater than 300 mg/dL while being treated, or not on appropriate lipid-lowering therapy within 4 weeks of study entry
* Karnofsky score <70%
* Prior history of allergy to sirolimus
* Requires voriconazole at time of study entry
* Currently receiving another investigational drug unless cleared by the principal investigator and sponsor
* Patients receiving BuCy as conditioning therapy

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-09; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is grade II-IV acute GVHD | One year

SECONDARY OUTCOMES:
Relapse-free survival | 2 years
Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olle Ringden, M.D. Ph.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Torlen J, Gaballa A, Remberger M, Mork LM, Sundberg B, Mattsson J, Uhlin M. Effect of Graft-versus-Host Disease Prophylaxis Regimens on T and B Cell Reconstitution after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2019 Jun;25(6):1260-1268. doi: 10.1016/j.bbmt.2019.01.029. Epub 2019 Jan 30. PMID 30710687
- [Derived] Torlen J, Ringden O, Garming-Legert K, Ljungman P, Winiarski J, Remes K, Itala-Remes M, Remberger M, Mattsson J. A prospective randomized trial comparing cyclosporine/methotrexate and tacrolimus/sirolimus as graft-versus-host disease prophylaxis after allogeneic hematopoietic stem cell transplantation. Haematologica. 2016 Nov;101(11):1417-1425. doi: 10.3324/haematol.2016.149294. Epub 2016 Aug 4. PMID 27662016